CLINICAL TRIAL: NCT06159985
Title: Effect of Left Posterior Pericardiotomy for the Prevention of Postoperative Atrial Fibrillation in Coronary Artery Bypass Grafting: A Prospective Randomized Controlled Trial
Brief Title: Effect of Left Posterior Pericardiotomy for the Prevention of POAF
Acronym: ELIMINATE-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Young Hwang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2309-096-1469
Record Dates: First submitted 2023-11-24; First posted 2023-12-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation New Onset; Pericardial Effusion
MeSH Terms: conditions — Coronary Artery Disease; Pericardial Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pericardiostomy (Active Comparator): The patients who were created with left posterior pericardiotomy during the operation
  Interventions: Procedure: left posterior pericardiostomy
- No pericardiostomy (No Intervention): The patients who were not created with left posterior pericardiotomy during the operation

INTERVENTIONS:
Procedure: left posterior pericardiostomy — In patients assigned to the study group, a 4-5 cm vertical incision posterior to the phrenic nerve and extending from the left inferior pulmonary vein to the diaphragm is performed.
  Arms: Pericardiostomy

SUMMARY:
This study is planned to evaluate the effect of left posterior pericardiotomy for the prevention of postoperative atrial fibrillation after coronary artery bypass grafting. Eligible patients will be randomized to be created or not to be created the left posterior pericardiotomy at the end of the operation, and the incidence of postoperative atrial fibrillation will be compared.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a common complication after cardiac surgery, particularly after coronary artery bypass grafting (CABG), and is associated with prolonged in-hospital stay and increased adverse outcomes, including death and stroke. There is evidence that pericardial effusion can trigger the occurence of POAF. Therefore, this study is aimed to evaluate the effect of left posterior pericardiotomy for the prevention of POAF after CABG.

Patients who are planned to undergo off-pump CABG will be randomized to be created or not to be created the left posterior pericardiotomy at the end of the operation, and the incidence of postoperative atrial fibrillation will be compared as the primary outcome. Secondary outcomes will include early clinical outcomes and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients who are planned to undergo coronary artery bypass grafting
* patients aged ≥19 years

Exclusion Criteria:

* patients who are planned to undergo other concomitant cardiac procedures (e.g. valve procedures, aorta procedures)
* patients who undergo coronary artery bypass grafting using cardiopulmonary bypass
* patients who are documented with paroxysmal, persistent, or permanent atrial fibrillation before operation
* patients who have a history of cardiac surgery
* patients who have a history of pericardial disease
* patients who have severe adhesion at left pleural cavity which precludes effective left posterior pericardiostomy
* patients who refuse to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
occurence rate of postoperative atrial fibrillation | From date of operation until postoperative day 7
  any short run of atrial fibrillation which occurred during postoperative period before discharge

SECONDARY OUTCOMES:
operative mortality | at 30 days
  death occurred during the index admission or within 30 days after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) and related data dictionaries available.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication
Access Criteria: IPD will be shared on reasonable request to the corresponding author.